CLINICAL TRIAL: NCT06508229
Title: Adebrelimab Combined With Albumin Paclitaxel and Nedaplatin as Neoadjuvant Therapy for Locally Advanced Resectable Esophageal Squamous Cell Carcinoma：a Prospective, Single Arm, Phase 2 Clinical Study
Brief Title: Adebrelimab Combined With Albumin Paclitaxel and Nedaplatin as Neoadjuvant Therapy for Locally Advanced Resectable ESCC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Jianqun Ma, MD, Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1316-HLJ-005
Record Dates: First submitted 2024-05-27; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: Adebrelimab; Chemotherapy; locally advanced ESCC
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — nedaplatin; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Immuno-chemotherapy for locally advanced ESCC (Experimental): Adebrelimab + albumin paclitaxel + nedaplatin
  Interventions: Drug: Adebrelimab; Drug: albumin paclitaxel; Drug: Nedaplatin

INTERVENTIONS:
Drug: Adebrelimab — adebrelimab, IV
  Other Names: SHR-1316
Drug: albumin paclitaxel — albumin paclitaxel, iv
  Other Names: Injectable paclitaxel (albumin bound)
Drug: Nedaplatin — Nedaplatin，IV
  Other Names: Nedaplatin for injection

SUMMARY:
This is a multi-center, single-arm, phase II clinical study designed to observe and evaluate the effectiveness and safety of adebrelimab combined with albumin paclitaxel and nedaplatin as neoadjuvant therapy for locally advanced resectable esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This study plans to include 65 patients who received 3 cycles of neoadjuvant therapy (Adebrelimab + albumin paclitaxel + nedaplatin) , and underwent surgery after the treatment was completed. The purpose of this study is to explore and evaluate the effectiveness and safety of adebrelimab combined with albumin paclitaxel and nedaplatin as neoadjuvant therapy for locally advanced resectable esophageal squamous cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 75 years old, no limit to male or female;
2. Surgically resectable locally advanced esophageal squamous cell carcinoma confirmed by histology or cytology (clinical stage: stage IIa-IIIb);
3. Have measurable lesions and meet RECIST v1.1) standards;
4. Have not received any anti-tumor systemic treatment for esophageal cancer in the past;
5. ECOG PS: 0-1 points;
6. Expected survival ≥12 weeks;
7. The functions of vital organs meet the following requirements:

   1. Routine blood examination (no blood transfusion within 14 days, no correction with hematopoietic stimulating factor drugs):Hemoglobin (Hb) ≥90 g/L; absolute neutrophil count (ANC) ≥1.5×109/L; platelets (PLT) ≥100×109/L; white blood cell count (WBC) ≥3.0×109/L;
   2. Biochemical examination: Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN; serum total bilirubin (TBIL) ≤1.5×ULN (Gilbert syndrome subjects, ≤ 3×ULN); serum creatinine (Cr) ≤1.5 ×ULN or creatinine clearance ≥50ml/min;
   3. Coagulation function: Activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤1.5×ULN;
   4. Doppler ultrasound evaluation: Left ventricular ejection fraction (LVEF) ≥50%;
8. Non-surgical sterilization or female patients of childbearing age need to use a medically approved contraceptive method during the study treatment period and within 3 months after the end of the study treatment period; female patients of childbearing age who have non-surgical sterilization must use a medically approved contraceptive method before study enrollment. The serum or urine HCG test must be negative within 72 hours; and must be non-lactating; for males, they should be surgically sterilized, or agree to use appropriate contraceptive methods during the trial and within 3 months after the last administration of the trial drug;
9. The patient voluntarily joined this study, signed the informed consent form (ICF), had good compliance, and cooperated with the follow-up.

Exclusion Criteria:

1. Patients with locked lymph node metastasis;
2. Have a history of other malignant tumors in the past 5 years, except for cervical carcinoma in situ or cutaneous squamous cell carcinoma that has been fully treated, or basal cell carcinoma of the skin that has been basically controlled;
3. Suffering from bleeding disorders or a history of bleeding disorders;
4. Have undergone major surgery or serious trauma within 4 weeks before taking the study drug for the first time;
5. Those with uncontrolled, symptomatic brain metastases or a history of uncontrollable mental illness or severe intellectual or cognitive dysfunction;
6. Have a history of interstitial lung disease and non-infectious pneumonia;
7. Suffering from active autoimmune diseases or a history of autoimmune diseases, such as interstitial pneumonia, colitis, hepatitis, hypophysitis, vasculitis, nephritis, hyperthyroidism, or reduced thyroid function after thyroid hormone replacement therapy can be included;
8. Have a history of immunodeficiency, including testing positive for HIV, suffering from other acquired or congenital immunodeficiency diseases, or a history of organ transplantation and allogeneic bone marrow transplantation;
9. Subjects have cardiovascular clinical symptoms or diseases that cannot be well controlled, including but not limited to:

1) NYHA class II or above heart failure; 2) Unstable angina; 3) Myocardial infarction within 1 year; 4) Clinically significant supraventricular or ventricular arrhythmia requiring clinical intervention; 10. Severe active infection requiring intravenous antibiotic treatment occurs within 4 weeks before using the study drug; 11. Those who are allergic to experimental drugs; 12. Patients who cannot comply with the trial protocol or cannot cooperate with follow-up visits; 13. Those who the researcher believes are not suitable to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2027-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
pathological complete remission rate | up to 24 months
  After neoadjuvant therapy and surgery, there were no residual surviving tumor cells in the tumor bed in the postoperative specimens (% RVT=0)

SECONDARY OUTCOMES:
R0 resection rate | up to 24 months
  The tumor lesion was completely removed, and no residual cancer cells were found on the cutting edge under the microscope
Main pathological remission | up to 24 months
  After neoadjuvant therapy and surgery, the proportion of tumor cells remaining alive in the tumor bed in the postoperative specimen is less than or equal to 10% (% RVT ≤ 10)
objective response rate | up to 24 months
  The proportion of patients whose tumors have shrunk to a certain amount and remained in remission for a certain period of time, including complete response (CR) and partial response (PR).
Disease-free survival | up to 24 months
  It was calculated from the time of first administration of study drug until disease progression or death.
overall survival | up to 24 months
  The time is calculated from the first administration of the study drug until death due to any cause (patients who were lost to follow-up are the last follow-up time; patients who are still alive at the end of the study are the end of follow-up date).
Number of participants with treatment related adverse events asassessed by CTCAE v5.0 | up to 24 months
  Proportion of patients with treatment-related adverse events recorded using CTCAE 5.0 criteria
Changes in the patient's mood | up to 24 months
  Use PHQ-9 and GAD-7 to record the changes in patients' emotions during treatment
The patient's nutritional status | up to 24 months
  Use PNI, CNI and mCONUT scoring standards to record changes in the patient's nutritional status during treatment
The pain level of patients | up to 24 months
  NRS and VAS pain rating scales were used to assess changes in patients' pain levels during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jianqun Ma, MD, Principal Investigator — Harbin Medical University Affiliated Cancer Hospital

IPD SHARING:
Plan to Share IPD: No